CLINICAL TRIAL: NCT07236216
Title: Effects of Transcranial Electrical Stimulation (tES) Combined With Cognitive-motor Dual-task Gait Training on Cortical Activity, Spinal Motoneuron Excitability, Cognition and Motor Performance in Stroke Individuals
Brief Title: Effects of tES Combined With CMDT Gait Training on Cognition, Cortical Activity, Spinal Motoneuron Excitability and Motor Performance in Stroke Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MU-CIRB 2025/304.1106
Record Dates: First submitted 2025-09-24; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hemorrhagic Stroke; Ischemic Stroke; Subacute Stroke; Chronic Stroke Patient
Keywords: stroke; electroencephalography; functional near infrared spectroscopy; event related potentials; rehabilitation; gait training; High-definition transcranial electrical stimulation
MeSH Terms: conditions — Hemorrhagic Stroke; Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active HD-tDCS with conventional physical therapy and CMDT gait training (Experimental): Participants will receive active tDCS for 20 minutes prior conventional physical therapy and CMDT gait training. They will be receive this intervention for 12 sessions (3 days/week for 4 weeks).
  Interventions: Device: High-definition transcranial direct current stimulation (Active); Other: Cognitive-motor dual task gait training; Other: Conventional Physical therapy
- Active HD-tACS with conventional physical therapy and CMDT gait training (Experimental): Participants will receive active tACS for 20 minutes prior conventional physical therapy and CMDT gait training. They will received this intervention for 12 sessions (3 days/week for 4 weeks).
  Interventions: Device: High-definition transcranial alternating stimulation (Active); Other: Cognitive-motor dual task gait training; Other: Conventional Physical therapy
- Sham stimulation witn conventional physical therapy and CMDT gait training (Sham Comparator): Participants will receive sham stimulation for 30 minutes prior conventional physical therapy and CMDT gait training. They will received this intervention for 12 sessions (3 days/week for 4 weeks).
  Interventions: Device: High-definition transcranial electrical stimulation (sham); Other: Cognitive-motor dual task gait training; Other: Conventional Physical therapy

INTERVENTIONS:
Device: High-definition transcranial direct current stimulation (Active) — Electrode placement based on the international 10-20 electroencephalography electrode system. The electrode will be place over ipsilesional hemisphere on the primary motor cortex area. Anodal electrode will be placed over C3 or C4, while other 4 return electrodes will be placed over FC1/FC2, FC5/FC6, CP1/CP2, CP5/CP6. Participants will be asked to sit comfortably during stimulation. Participants will receive active HD-tDCS with intensity 2.0 mA for 20 minutes with 30-sec ramp-up and ramp-down.
  Other Names: HD-tDCS; starstim; Neuroelectrics, Spain
  Arms: Active HD-tDCS with conventional physical therapy and CMDT gait training
Device: High-definition transcranial alternating stimulation (Active) — Electrode placement based on the international 10-20 electroencephalography electrode system. The electrode will be place over ipsilesional hemisphere on the primary motor cortex area. Anodal electrode will be placed over C3 or C4, while other 4 return electrodes will be placed over FC1/FC2, FC5/FC6, CP1/CP2, CP5/CP6. Participants will be asked to sit comfortably during stimulation. Participants will receive active HD-tACS with intensity 2.0 mA for 20 minutes with frequency 70 Hz.
  Other Names: HD-tACS; starstim; Neuroelectrics, Spian
  Arms: Active HD-tACS with conventional physical therapy and CMDT gait training
Device: High-definition transcranial electrical stimulation (sham) — Electrode placement based on the international 10-20 electroencephalography electrode system. The electrode will be place over ipsilesional hemisphere on the primary motor cortex area. Anodal electrode will be placed over C3 or C4, while other 4 return electrodes will be placed over FC1/FC2, FC5/FC6, CP1/CP2, CP5/CP6. Participants will be asked to sit comfortably during stimulation. Participants will receive active HD-tDCS with intensity 2.0 mA for 20 minutes with electrical current flows 1-minute, with 30-second ramp-up and ramp-down, and no electrical current flow after first 1 minute to the end of stimulation.
  Other Names: Sham stimulation; starstim; Neuroelectrics, Spian
  Arms: Sham stimulation witn conventional physical therapy and CMDT gait training
Other: Cognitive-motor dual task gait training — Participants will be trained in cognitive-motor dual task gait training by using Zebris Rehawalk gait analysis and gait training. Participants will be asked to walk on treadmill while response to cognitive tasks on the computer screen, which is placed in front of participants. Treadmill speed will be set according to participants' preferred speed. Cognitive tasks involve color tasks and math tasks.
Other: Conventional Physical therapy — Conventional physical therapy starts immediately after stimulation ends. In 1-hour of conventional physical therapy involving 10 minutes of upper and lower extremity stretching, 20 minutes of upper extremity training, and 30 minutes of lower extremity training.

SUMMARY:
The present study will use transcranial electrical stimulation (tES) which are transcranial direct current stimulation (tDCS) and transcranial alternating current stimulation (tACS) combined with conventional physical therapy and cognitive-motor dual task gait training in sub-acute (at least 2 weeks after stroke onset) to chronic (within 5 years post-stroke) to investigate the effect on cortical activity, spinal motoneuron excitability, cognition and motor performance. The findings may enhance the evidence to support usages of tES for improvimg cognition, motor performance as well as cortical activity and spinal motoneuron excitability in a clinical setting.

DETAILED DESCRIPTION:
Stroke is a sudden neurological event which is leading cause of death and disability. An impaired blood flow and oxygen supply leading to neuronal cell death follwoing stroke. In addition, an electroencephalography demonstrated a decrease of high frequency power bands (alpha and beta) and increase of low frequency bands (theta and delta). An increase in delta frequency is negatively correlated with cognition, while an increase in high-frequency bands are correlatedw ith an improvement of motor recovery and cognition. Furthermore, functional near-infrared spectroscopy (fNIRS) which is a non-invasive neuroimaging can monitors improvements in cortical activity throughchanges in cerebral blood flow and oxygen consumptions.

Follwoing stroke, an alterations of cortical activity between ipsileasional hemisphere and contralesion hemisphere affect the spinal lelvel as it leads to increase spinal motoneuron excitability. An increase of spinal motoneuron excitability is likely due to abnormal control from cortex to spinal cord via descending pathway. Furthermore, hyperexcitability of spinal motoneuron is associated with post-stroke spasticity. However, the excat mechanisms of spasticity in post stroke remians unclear. Potential causes include imbalance in descending pathway regulation, abnormal intraspinal processing, and altered muscular viscoelasticity. Changes in spinal motoneuron excitability can be assessed using Hoffmann's reflex (H-reflex).

Motor imapirments following stroke affects activities of daily living (ADLs), moreover cognitive impairements is commonly obsrved in post-stroke individuals that may limits motor and functional recovery and limits effectiveness of rehabilitation. These impairments affect both single- and duals-task activities, especially walking performance and increasing risk of falls in stroke individuals. In recent years, combining bottom-up and top-down approaches has been greater potential in promoting neural plasticity and enhancing motor recovery compared to single approach. Bottom-up approaches refers to rehabilitation that act on physical level and expected chnages in nervous system level, while top-down approach induce change in cortical level to induce change in motor function or physical level. The non-invasive brain stimulation (NIBS) is a top-down approach that enhance neural plasticity and mediated motor-relearning in neurological conditions. Transcranial electrical stimulation (tES) is one of NIBS which the most coom tES techniques are transcranial direct current stimulation (tDCS) and transcranial alternating currnt stimulation (tACS). Both tDCS and tACS are different in their wave forms. tDCS delivers a weak direct current with polartiy-specific effects, while tACS enhance neural plasticity and endogenous brain wave with frequency-specific. A recent review demonstrated the effectiveness of tDCS in improvement of motor function, functional abilities and cognitive function. Furthermore, a previous study demonstrated an improvement in cognitive function and ADLs following combining 2mA of tDCS with CMDT training. However, the amount of evidence on the effects of tACS is much less than that for tDCS, as it has only recently started to gain interest. The frequency used in tACS study mainly follows the association of brain wave and function. A previous review showed that gamma tACS enhance cognitive performance, working memory and logical thinking. In healthy population, a previous study demonstrated that applied gamma-tACS over M1 significantly improved velocity and acceleration of visuomotor task; nevertheless, this improvement did not found in beta-tACS. To provide evidence of the effects of tACS in the stroke population and to identify which type of transcranial electrical stimulation is most appropriate for stroke rehabilitation, a comparison between tDCS and tACS is necessary. Both tES technique will be combined with conventional physical therapy for 12 sessions (3 days/week for 4 weeks). tES will be provided for 20 minutes, then followed by convention physical therapy (1-hour) and cognitive-motor dual-task gait training (30-minute). Cortical activity will be assessed by EEG and fNIRS. Absoule spectral power of each frequency bands (alpha, beta, delta, and theta) will be analyze. The hemodynamics data will be analyze to represent changes of blood flow to the brain after intervention. The Hmax/Mmax ratio from flexor carpi radialis and soleus will be recorded to represent changes in spinal motoneuron excitability. The Fugl-Meyer assessment of upper and lower extremity and Timed up and go will be used to represent clinical outcomes of motor function and performance. The ERP recorded during Stroop color and word test and 2-Back test will be assessed together with the Montreal Cognitive Assessment (MoCA) in Thai version. Furthermore, behavoral data i.e. response time, accuracy will be collected to analyse to represent cogniton. For walking performance, dual-task interference or dual-task costs will be employed from dual-task walking. All outcomes will be assessed at baseline, post-intervention, 1-month follow-up, and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral stroke individuals aged 18-80 years.
2. A first-ever stroke.
3. Stroke onset from at least 2 weeks-5 years.
4. Able to walk independently with or without gait aids (modified Rankin scale (mRS) 1-3)
5. Montreal cognitive Assessment-Thai version (MoCA-T) greater than or equal to 20 scores.
6. Ability to read, communicate, follow and understand instructions.

Exclusion Criteria:

1. Presence of any psychological or neurological antecedent, unstable medical conditions or condition that may increase risk of stimulation such as epilepsy, seizure, and history of brain injury
2. Having unstable cardiovascular disease or respiratory disease, and uncontrolled chronic disease such as diabetes mellitus (DM), hypertension (HT) and chronic kidney disease (CKD)
3. Receiving other non-invasive brain stimulation or additional intervention such as TMS, PMS or acupuncture
4. Presence of metal implantation, intracranial shunt, cochlear implantation, or cardiac pacemakers.
5. Presence of an opened wound, infectious wound around scalp or craniectomy with unreplaced bone flap
6. Moderate pain (numeric pain rating score > 4/10) in any joint of the upper or lower limb, whether paretic or non-paretic
7. Presence of color blindness
8. Presence of any substance use including cannabis and kratom

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Absolute power | Baseline, 1-day post-intervention, 1-month follow-up and 3-month follow-up
  The raw data from electroencephalographyt (EEG) in 5-min of eye-open and eye-close conditions converted to the power distribution of brain waves in different frequencies (i.e. delta, theta, and beta) usign a Fast Fourier Transformation (FFT)

SECONDARY OUTCOMES:
Blood oxygenation level | Baseline, 1-day post-intervention, 1-moth follow-up and 3-month follow-up
  Changes in concentration of hemoglobin between oxygenated hemoglobin (HbO2) and deoxygenated hemoglobin (HbR) in the brain, which can indicate brain function in different areas are assessed by Functional Near-Infrared Spectroscopy (fNIRS)
Event Related Potential (ERP) | Baseline, 1-day post-intervention, 1-month follow-up and 3-month follow-up
  ERP is a non-invasive measurement tool that detects a very small voltage generated by brain activity in response to a specific event (i.e. Stroop test, N-back test). This is a signal averaging form of EEG that detects signals starting from the onset of a stimulus to evaluate brain responses over time, those occurring at 200 milliseconds (P200), or 300 milliseconds (P300) .
Fugl-Meyer assessment (FMA) of upper and lower extremities | Baseline, 1-day post-intervention, 1-month follow-up, and 3-month follow-up
  The FMA is a clinical assessment that quantified level of motor impairement and evaluate recovery in post-stroke. The FMA Includes 33 items for the upper extremity and 17 items for the lower extremity, totaling 100 points. Higher scores indicate better motor performance.
Montreal Cognitive Assessment | Baseline, 1-day post-intervention, 1-month follow-up and 3-month follow-up
  The Montreal Cognitive Assessment (MoCA) is used to assess cognitive functioning in eight domains: Visuospatial and executive function, Naming, Attention, Language, Abstraction, Delayed recall, Orientation, Short-term memory. Participants are instructed to complete both paper-based and verbal question-answering activities, such as drawing pictures, sorting numbers, naming animals, and reviewing vocabulary. The maximum total score is 30 points, with a high score indicating a good level of cognitive.
Timed up and go test | Baseline, 1-day post-intervention, 1-month follow-up and 3-month follow-up
  Participants wear regular footware and if they have normally used gait aid, it is allowed to use in the test. The test measures the time taken when the participants stand up from the chair, walk at normal pace for 3 meters, turn around, walk back for 3 meters, and then sit on a chair.
Cognitive-motor interference (CMI) | Baseline, 1-day post-intervention, 1-month follow-up and 3-month follow-up
  CMI refers to a decline in performance observed when a person simultaneously performs a cognitive and motor task, compared to performing a single- or dual-task separately. Managing both tasks requires divided attention, and interference arises when these cognitive resources are insufficient to maintain performance in both domains. The CMI can be quantified by the dual-task cost (DTC). The DTC is calculated by comparing the performance difference between single-task and dual-task conditions. Participants will be asked to perform 2 walking conditions on the treadmill (Zebris Rehawalk gait analysis and gait training). The walking conditions are single-walking and cognitive-motor dual task walking (CMDT walking). For single-walking, participants will be asked to walk at their preferred speed. For CMDT walking, participants will walk and response to stimuli on the screen simultaneously. During the test, stride length, step length, cadence and accuracy of response
Soleus H-reflex | Baseline, 1-day post-intervention, 1-month follow-up and 3-month follow-up
  The H-reflex is an electrophysiological measurement used to assess spinal excitability. For the soleus H-reflex , participants will be in prone position with ankle in neutral position. A bipolar electrode will be placed over the popliteal fossa, and the surface EMG electrode will be attached to the motor point of the soleus muscle (two electrodes on the lower 1/3 of the lower leg), and the lateral malleolus (ground electrode).
  The electrical stimulation starts at a minimal intensity, increasing until an H-reflex response is detected, continuing to supramaximal intensity to elicit an M-wave. H-reflex latency, maximum H- and M-wave responses will be recorded. The Hmax/Mmax ratio will be calculated from maximum H- and M-wave amplitude responses.
Flexor carpi radialis (FCR) H-reflexe | Baseline, 1-day post-intervention, 1-month follow-up and 3-month follow-up
  For the FCR H-reflex, participants will sit with their wrist in neutral, forearm mid-pronated, and their elbow flexed at 45 degrees, with slight shoulder abduction, flexion, and neutral rotation (68). Bipolar electrode will be placed medially to cubital fossa and the biceps brachii tendon. Two surface electrodes will be positioned over the FCR (1/3 of the distance from the medial epicondyle to the radial styloid), with a grounded electrode placed over radial styloid process. For the FCR H-reflex (Figure 10), participants will sit with their wrist in neutral, forearm mid-pronated, and their elbow flexed at 45 degrees, with slight shoulder abduction, flexion, and neutral rotation (68). Bipolar electrode will be placed medially to cubital fossa and the biceps brachii tendon. Two surface electrodes will be positioned over the FCR (1/3 of the distance from the medial epicondyle to the radial styloid) (69), with a grounded electrode placed over radial styloid process.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No